CLINICAL TRIAL: NCT00215631
Title: Can Tadalafil (Cialis)® Maintain Erectile Function In Patients Treated With External-beam Radiotherapy For Prostate Cancer? A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Can Tadalafil Maintain Erectile Function In Patients Treated With Radiotherapy For Prostate Cancer?
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2004-165
Record Dates: First submitted 2005-09-18; First posted 2005-09-22 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2007-04

CONDITIONS: Prostate Cancer; Erectile Dysfunction
Keywords: prostate cancer; radiotherapy; erectile dysfunction; tadalafil
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Tadalafil

INTERVENTIONS:
Drug: tadalafil

SUMMARY:
Because of the high incidence of post-radiation erectile dysfunction (ED), up to 72% after external-beam radiotherapy, this patient category represents a most difficult therapeutic challenge. Therefore, prevention of ED could be more effective than treatment. Tadalafil, a new phosphodiesterase type 5 inhibitor, has been recently introduced. No studies have investigated the efficacy of tadalafil in preventing ED in patients undergoing radiotherapy for prostate cancer. Efficacy of tadalafil can last up to 36 hours after intake. This will result in a prolonged and continuos enhancement of penile vascular responsiveness. This randomized, double-blind, placebo-controlled study has been designed to evaluate the efficacy of 20-mg of tadalafil administered for 12 months in maintaining erectile function of potent patients undergoing external-beam radiotherapy for prostate cancer.

DETAILED DESCRIPTION:
It will be a double-blind, placebo-controlled, randomized trial. Patients scheduled for external-beam radiotherapy for prostate cancer will start using tadalafil 20 mg or placebo the first day of radiation. The blinded medication (active drug or placebo) has to be taken once every two days starting the day of the first radiation up to 12 months (52 weeks) after radiotherapy. The active drug or placebo may be taken at bedtime unrelated to sexual activity. In case of side effects the dose can be reduced to 10 mg. Erectile function will be assessed every 3 months up to 6 weeks (week 58) after discontinuation of drug treatment by using questions 3 and 4 of the International Index of Erectile Function (IIEF). Responders (maintained erectile function) are defined as having a combined score of >=8 for the IIEF questions 3 and 4.

ELIGIBILITY:
Inclusion Criteria:

1. Men, at least 18 years of age, willing to participate in the study and willing to regularly attempt sexual activity.
2. Patients with histologically proven prostate cancer.
3. Provide signed informed consent.
4. Patients with normal erectile function defined as a combined score >=8 of questions 3 and 4 of the IIEF.
5. Agree not to use any other ED treatment during the study.

Exclusion Criteria:

1. Use of any treatment for ED before the start of the study.
2. History of pelvic surgery (including radical prostatectomy)
3. History of penile implant
4. The presence of penile deformity that makes sexual intercourse difficult or impossible.
5. Patients with chronic stable angina treated with long-acting nitrates, or patients with chronic stable angina who have required short-acting nitrates in the last 90 days, or angina occurring during sexual intercourse in the last 6 months.
6. Patients with unstable angina, history of myocardial infarction or coronary artery bypass graft surgery or percutaneous coronary intervention (eg, angioplasty or stent placement) within 90 days before screening.
7. Any supraventricular arrhythmia with an uncontrolled ventricular response (mean heart rate >100 bpm) at rest despite medical or device therapy, or any history of spontaneous or induced sustained ventricular tachycardia (heart rate >100 bpm for 30 sec) despite medical or device therapy, or the presence of an automatic internal cardioverter-defibrillator.
8. A history of sudden cardiac arrest despite medical or device therapy.
9. Any evidence of congestive heart failure or a new, significant conduction defect within 90 days before screening.
10. Systolic blood pressure >170 or <90 mm Hg or diastolic blood pressure >100 or <50 mm Hg, or patients with a history of malignant hypertension.
11. History of significant central nervous system injuries (including stroke and spinal cord injury) within the 6 months before screening.
12. History of HIV infection.
13. Any condition that would interfere with the patient's ability to provide informed consent or comply with study instructions, would place patient at increased risk, or might confound the interpretation of the study results.
14. Treatment with cancer chemotherapy.
15. History of drug, alcohol, or substance abuse within the 6 months before screening.
16. Have any condition, limitation, or disease that could, in the judgment of the investigator, preclude evaluation of response to tadalafil.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-10; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy, and safety, of 20 mg tadalafil once every 2 days, in comparison with placebo, to maintain erectile function of patients undergoing external-beam radiotherapy for prostate cancer.

SECONDARY OUTCOMES:
Erectile function defined as the sum of questions 3 and 4 of the IIEF questionnaire every 3 months till the end of the study (at 3-6-12-24 months).
Erectile function domain of the IIEF, defined as the sum of questions 1-5, and 15 of the IIEF questionnaire, questions 2 and 3 of the Sexual Encounter Profile (SEP), and responses to the other questions of the IIEF, at 3-6-12-24 months after initiation

CONTACTS AND LOCATIONS:
Overall Officials: Luca Incrocci, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC-Daniel den Hoed Cancer, Rotterdam, Netherlands